CLINICAL TRIAL: NCT02990403
Title: The Novel Immunomodulatory and Anticoagulant Therapies for Recurrent Pregnancy Loss
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Shihua Bao, Principal Investigator, Shanghai First Maternity and Infant Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiFMIH-0003
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2016-12

CONDITIONS: Recurrent Pregnancy Loss
MeSH Terms: interventions — Aspirin; Heparin; Prednisone; Immunoglobulins; Dydrogesterone

ARMS (5):
- aspirin+LMWH group (Experimental): aspirin, 75-100mg/day, po,bid + low molecular weight heparin,4100U,hypodermic injection，qd
  Interventions: Drug: Aspirin; Drug: Heparin
- aspirin+LMWH+immunoglobulin group (Experimental): aspirin, 75-100mg/day, po,bid + low molecular weight heparin,4100IU/day,hypodermic injection,qd + immunoglobulin 300mg/kg（with 100ml normal saline）,intravenous injection,once every two weeks
  Interventions: Drug: Aspirin; Drug: Heparin; Drug: Immunoglobulin
- aspirin+LMWH+prednisone group (Experimental): aspirin, 75-100mg/day, po,bid + low molecular weight heparin,4100IU/day,hypodermic injection,qd + prednisone,5-10mg/day,po,qd
  Interventions: Drug: Aspirin; Drug: Heparin; Drug: Prednisone
- aspirin+LMWH+IVIG+prednisone group (Experimental): aspirin, 75-100mg/day, po,bid + low molecular weight heparin,4100IU/day,hypodermic injection,qd + immunoglobulin 300mg/kg（with 100ml normal saline）,intravenous injection,once every two weeks + prednisone,5-10mg/day,po,qd
  Interventions: Drug: Aspirin; Drug: Heparin; Drug: Prednisone; Drug: Immunoglobulin
- dydrogesterone group (Other): dydrogesterone 20-30mg/day, po, tid
  Interventions: Drug: Dydrogesterone

INTERVENTIONS:
Drug: Aspirin
  Arms: aspirin+LMWH group; aspirin+LMWH+IVIG+prednisone group; aspirin+LMWH+immunoglobulin group; aspirin+LMWH+prednisone group
Drug: Heparin
  Arms: aspirin+LMWH group; aspirin+LMWH+IVIG+prednisone group; aspirin+LMWH+immunoglobulin group; aspirin+LMWH+prednisone group
Drug: Prednisone
  Arms: aspirin+LMWH+IVIG+prednisone group; aspirin+LMWH+prednisone group
Drug: Immunoglobulin
  Arms: aspirin+LMWH+IVIG+prednisone group; aspirin+LMWH+immunoglobulin group
Drug: Dydrogesterone
  Arms: dydrogesterone group

SUMMARY:
In this clinical cohort study, the investigators are going to observe the efficacy of anti-coagulation and immune therapy in the treatment of recurrent pregnancy loss with a prospective randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

- Woman who had 2 miscarriage before 12(th) week of gestation.The patient who is diagnosed as thrombophilia with recurrent pregnancy loss. Signed consent form.

Exclusion Criteria:

1. having experienced severe allergies, trauma history and/or operation history within 3 months.
2. with a history of mental illness and/or family history of mental illness limb disabled.
3. taking medicine within one month.
4. suffering major events or having mood swings.
5. having internal and surgical disease(after having variety of physical examination such as electrocardiogram/hepatic and renal function/blood routine and urine routine)
6. chromosome aberrations in anyone of the couple.
7. patients who have drugs contraindications

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-06-10 (Estimated); Study Completion 2018-12-22 (Estimated)

PRIMARY OUTCOMES:
live birth | through study completion, an average of 3 year
  live birth means success pregnancy（more than gestational age of 20 weeks）

SECONDARY OUTCOMES:
D-dimer | through study completion, an average of 3 year
Uterine artery blood flow | through study completion, an average of 3 year
human chorionic gonadotropin | through study completion, an average of 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai first Maternity and Infant health hospital, Tong Ji University, Shanghai, China